CLINICAL TRIAL: NCT03977987
Title: Maternal Nucleos(t)Ide Analogue Use and Infants Immunoprophylaxis to Eliminate Hepatitis B Infection in the Real World Setting
Brief Title: Maternal Antiviral Treatment and Infants Immunoprophylaxis in the Prevention of Mother-to-child Transmission
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Other Study IDs: RWD-0
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Hepatitis B
Keywords: hepatitis B; mother-to-children transmission; antiviral treatment; immunoprophylaxis
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The treatment group: Pregnant women with high HBV DNA level > 2*10^6 IU/ml who agree to receive the antiviral treatment during the late pregnancy.
  Interventions: Drug: nucleos(t)ide analogue
- The control group with high HBV DNA level: Pregnant women with high HBV DNA level > 2*10^6 IU/ml who decline to receive the antiviral treatment during the late pregnancy.
- The control group with low HBV DNA level: Pregnant women with high HBV DNA level < 2*10^6 IU/ml

INTERVENTIONS:
Drug: nucleos(t)ide analogue — Pregnant women in this group agree to receive nucleos(t)ide analogue (tenofovir or telbivudine) daily from the 28 weeks of pregnancy to delivery.
  Groups: The treatment group

SUMMARY:
The effective control of nucleos(t)ide analogues for patients infected with hepatitis B has significantly curbed the horizontal transmission of hepatitis B. However, the vertical transmission remains a serious threat to public health for directly increasing the burden of hepatitis B worldwide with the transmission rate up to 80 to 90% among high HBV DNA level if untreated. Currently, the effective prevention of mother-to-child transmission is credited to the implement of HBV vaccination and hepatitis B virus immunoglobin. To leave nobody behind, a growing body of evidence has been yielded to support the use of nucleos(t)ide analogues in the mothers during the late pregnancy. However, the clinical practice can be more complex. Therefore, investigators aim to assess the effectiveness of maternal antiviral therapy and different infants immunoprophylaxis strategy in the prevention of chronic hepatitis infection among children whose mothers were infected with chronic hepatitis B infection in the real world setting.

DETAILED DESCRIPTION:
From 2011 to 2017, the investigators consecutively enrolled the pregnant women with chronic hepatitis B infection who were less than 28 weeks pregnant and not treated with nucleos(t)ide analogues during pregnancy. The investigators recommended those pregnant women with HBV DNA > 2*10^6 IU/ml to receive nucleos(t)ide analogues from 28 weeks of pregnancy to delivery. Patients who agreed the antiviral treatment would assigned to the treatment group and those who declined it were assigned to the control group with high HBV DNA level. Meanwhile, those pregnant women with HBV DNA < 2*10^6 IU/ml was assigned as the control group with low HBV DNA level. All infants would be instructed to receive hepatitis B vaccine and hepatitis B virus immunoglobulin within 24 hours after birth, defined as the standard immunoprophylaxis strategy and encouraged to receive immunoprophylaxis within 2 hours after birth, defined as the aggressive immunoprophylaxis strategy. Umbilical cord blood were collected to determine the HBV serological markers and HBV DNA level. Children were followed every three to four years until December 2018.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive women who were less than 28 weeks pregnant and underwent routine testing for HBV at the Department of Infectious Diseases of Taicang First People's Hospital at least twice during pregnancy

Exclusion Criteria:

* women treated with antiviral drugs during pregnancy.
* drug hypersensitivity;
* abnormal renal laboratory results;
* coinfection with human immunodeficiency virus or other human hepatitis viruses.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the real-world setting, we recruited consecutively HBsAg positive women who were less than 28 weeks pregnant and underwent routine testing for HBV at the Department of Infectious Diseases of Taicang First People's Hospital at least twice during pregnancy. Patients were excluded from participation if they had been treated with antiviral drugs during pregnancy. Additional exclusion criteria were drug hypersensitivity, abnormal renal laboratory results, coinfection with human immunodeficiency virus or other human hepatitis viruses.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
The proportion of children who developed chronic HBV infection between the treatment group and two control groups in the real-world setting. | December, 2018
  We compare the proportion of children with chronic HBV born to mothers from three groups in the real life setting

SECONDARY OUTCOMES:
the proportion of children who developed chronic HBV infection between the treatment group and two control groups among infants who followed the standardized immunoprophylaxis strategy | December, 2018
  We compare the proportion of children with chronic HBV born to mothers from three groups who followed the standardized immunoprophylaxis strategy
the proportion of children who developed chronic HBV infection between the treatment group and two control groups among infants who followed the aggressive immunoprophylaxis strategy | December, 2018
  We compare the proportion of children with chronic HBV born to mothers from three groups who followed the aggressive immunoprophylaxis strategy
The proportion of children with detectable HBV DNA and HBsAg in umbilical cord blood | At delivery
  We compare the proportion of children with detectable HBV DNA and HBsAg in umbilical cord blood born to mothers from three groups
The HBV DNA level of mothers among three groups | Within one week before delivery.
  We compare the HBV DNA level of mothers among three groups within one week before delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Yonglan Pu, Study Director — The First People's Hospital of Taicang
Locations (1):
- The First People's Hospital of Taicang, Suzhou, Jiangsu, China